CLINICAL TRIAL: NCT05903144
Title: Influence of Manual Diaphragm Release Combined With Conventional Breathing Exercises and Prone Positioning on Pulmonary Functions in Women With COVID-19
Brief Title: Influence of Manual Diaphragm Release on Pulmonary Functions in Women With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mona abd el raouf ghallab, lecturer at faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PFT in COVID-19
Record Dates: First submitted 2023-06-09; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: COVID-19 Pneumonia
Keywords: Breathing Exercise; COVID-19; manual diaphragmatic release; Pulmonary function parameters
MeSH Terms: conditions — COVID-19 | interventions — Musculoskeletal Manipulations; Breathing Exercises; Prone Position

STUDY DESIGN:
Intervention Model Description: Forty females were randomly assigned to two groups. Group A received manual diaphragm release with conventional breathing exercises and prone positioning. Group B received conventional breathing exercises and prone positioning. Both groups took their prescribed medications. Their ages ranged from 35 to 45 years and with moderate COVID-19 illness. Any cases with mild and severe COVID-19 illness, ICU admission, and chest diseases were excluded.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): they received manual diaphragm release with conventional breathing exercises and prone positioning in addition to their prescribed medications.
  Interventions: Other: manual therapy; Other: breathing exercise and prone position alone
- Control group (Active Comparator): they received conventional breathing exercises and prone positioning alone in addition to their prescribed medications.
  Interventions: Other: breathing exercise and prone position alone

INTERVENTIONS:
Other: manual therapy — manual diaphragmatic release technique combined with breathing exercise
  Arms: Study group
Other: breathing exercise and prone position alone — deep breathing exercise and prone position

SUMMARY:
Manual noninvasive respiratory techniques gained interest to treat respiratory pathologies related to COVID 19. This study designed to determine the combined effect of manual diaphragmatic release technique with the effect of conventional breathing exercises and prone positioning on pulmonary function parameters (FVC, FEV1, PEF, FEV1/FVC, FEF25, FEF50, FEF75, FEF25/75).

DETAILED DESCRIPTION:
Forty females were randomly assigned to two groups. Group A received manual diaphragm release with conventional breathing exercises and prone positioning. Group B received conventional breathing exercises and prone positioning. Both groups took their prescribed medications. Their ages ranged from 35 to 45 years and with moderate COVID-19 illness. Any cases with mild and severe COVID-19 illness, ICU admission, and chest diseases were excluded.

Main measures: pulmonary function parameters (FVC, FEV1, PEF, FEV1/FVC, FEF25, FEF50, FEF75, FEF25/75).

ELIGIBILITY:
Inclusion Criteria:

* women with moderate COVID-19 illness diagnosed by a physician.
* Patients with o2 saturation >94%Nonsmoker subjects.
* age ranging from 35-45 years.
* body mass index from 25 to 34 kg/m2.

Exclusion Criteria:

* Unstable hemodynamic status.
* Acute respiratory failure requiring intubation and impaired consciousness.
* Inability to collaborate with prone positioning with refusal.
* Change of mental status hindering response to instructions.
* Poorly controlled hypertension (Mean systolic BP > 140 mmhg and \or diastolic BP > 40 mmhg).
* Patients who take continuous o2 supplementation.
* Smoking.
* Other chest diseases as (COPD-asthma-tuberculosis-cancer).
* Male patients.

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
forced vital capacity FVC | pre study and 3 weeks post study for all participants
  the amount of air that can be forcibly exhaled from your lungs after taking the deepest breath possible which is a common breathing test to check lung function.
FEV1 | pre study and 3 weeks post study for all participants
  the maximum amount of air that the subject can forcibly expel during the first second following maximal inhalation
PEF | pre study and 3 weeks post study for all participants
  show the amount and rate of air that can be forcefully breathed out of the lungs.
FEV1/FVC | pre study and 3 weeks post study for all participants
  FEV1/FVC, also known as FEV1%) can help distinguish obstructive and restrictive lung diseases.
PEF25% | pre study and 3 weeks post study for all participants
  Peak expiratory flow at 25% of fvc and the most sensitive measure of airflow in peripheral airways where primary airflow obstruction originates.
PEF50% | pre study and 3 weeks post study for all participants
  Peak expiratory flow at 50% ofFVC
PEF 75% | pre study and 3 weeks post study for all participants
  Peak expiratory flow at 75% of FVC
PEF 25%/75% | pre study and 3 weeks post study for all participants
  Maximum flow rate in the middle 50% of forced expiration.

CONTACTS AND LOCATIONS:
Overall Officials: mona M ghallab, doctoral, Principal Investigator — PHD and lecturer of physical therapy for cardiovascular disease and geriatrics,cairo univeristy; neveen M nawar, master, Study Chair — master degree of physical therapy for cardiovascular disease and geriatrics, cairo univeristy; karim I safaan, doctoral, Study Director — PHD and lecturer of physical therapy for Surgery, cairo univeristy; kerolous I shehata, doctoral, Study Director — PHD and lecturer Department of women health/ faculty of physical therapy /cairo university; Amira I mostafa, doctoral, Study Director — PHD and Assistant professor of chest disease Faculty of medicine cairo univeristy; mona A mohamed, doctoral, Study Chair — PHD and lecturer of physical therapy for cardiovascular disease and geriatrics,cairo univeristy
Locations (1):
- Cairo Univeristy, Multiple Locations, Giza Governorate, Egypt

REFERENCES:
- [Background] Rocha T, Souza H, Brandao DC, Rattes C, Ribeiro L, Campos SL, Aliverti A, de Andrade AD. The Manual Diaphragm Release Technique improves diaphragmatic mobility, inspiratory capacity and exercise capacity in people with chronic obstructive pulmonary disease: a randomised trial. J Physiother. 2015 Oct;61(4):182-9. doi: 10.1016/j.jphys.2015.08.009. Epub 2015 Sep 19. PMID 26386894
- [Background] Ahmad AM, Nawar NM, Dabess HM, Gallab MA. Effect of diaphragm manual release versus conventional breathing exercises and prone positioning on physical functional performance in women with COVID-19: A randomized trial. J Bodyw Mov Ther. 2023 Jul;35:311-319. doi: 10.1016/j.jbmt.2023.04.064. Epub 2023 Apr 21. PMID 37330786
- [Background] Elnaggar RK, Shendy MA, Mahmoud MZ. Prospective Effects of Manual Diaphragmatic Release and Thoracic Lymphatic Pumping in Childhood Asthma. Respir Care. 2019 Nov;64(11):1422-1432. doi: 10.4187/respcare.06716. Epub 2019 Jul 23. PMID 31337743
- [Background] Gonzalez-Alvarez FJ, Valenza MC, Torres-Sanchez I, Cabrera-Martos I, Rodriguez-Torres J, Castellote-Caballero Y. Effects of diaphragm stretching on posterior chain muscle kinematics and rib cage and abdominal excursion: a randomized controlled trial. Braz J Phys Ther. 2016 Jun 16;20(5):405-411. doi: 10.1590/bjpt-rbf.2014.0169. PMID 27333481
- [Background] Courtney R., Biland G., Ryan A., et al. Improvements in multi-dimensional measures of dysfunctional breathing in asthma patients after a combined manual therapy and breathing retraining protocol: a case series report. International Journal of Osteopathic Medicine 2019: (31) 36-43.
- [Background] Nagy EN, Elimy DA, Ali AY, Ezzelregal HG, Elsayed MM. Influence of Manual Diaphragm Release Technique Combined with Inspiratory Muscle Training on Selected Persistent Symptoms in Men with Post-Covid-19 Syndrome: A Randomized Controlled Trial. J Rehabil Med. 2022 Oct 20;54:jrm00330. doi: 10.2340/jrm.v54.3972. PMID 36121338